CLINICAL TRIAL: NCT06082037
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase 3 Study, Followed by Open-label Extensions, to Evaluate the Efficacy of Oral Belumosudil in Adult Participants With Chronic Lung Allograft Dysfunction (CLAD) Following Bilateral Lung Transplantation
Brief Title: A Study to Test How Effective Belumosudil Tablets Are for Treating Adult Participants With Chronic Lung Allograft Dysfunction
Acronym: ROCKaspire
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Meiji Seika Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17801; U1111-1280-6777 (Registry Identifier: ICTRP); 2023-503462-23 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-10-07; First posted 2023-10-13 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Lung Transplant Rejection
MeSH Terms: interventions — belumosudil; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belumosudil + Azithromycin (Experimental): Participants will receive 200 mg belumosudil orally once daily
  Interventions: Drug: Belumosudil; Drug: Azithromycin
- Placebo + Azithromycin (Placebo Comparator): Participants will receive placebo orally once daily
  Interventions: Drug: Azithromycin; Drug: Placebo

INTERVENTIONS:
Drug: Belumosudil — Tablet, Oral
  Other Names: REZUROCK
  Arms: Belumosudil + Azithromycin
Drug: Azithromycin — Depends on pharmaceutical presentation, Oral
Drug: Placebo — Tablet, Oral
  Arms: Placebo + Azithromycin

SUMMARY:
This double-blind, randomized, placebo-controlled, multinational, multicenter, parallel-group, Phase 3, 2-arm, study will investigate the efficacy and safety of belumosudil compared with placebo, both administered on top of azithromycin and standard-of-care regimen of immunosuppression in male or female participants at least 1 year after bilateral lung transplant, who are at least 18 years of age and who have evidence of progressive CLAD despite azithromycin therapy.

Study details include:

The study duration will be up to 31 weeks for participants not entering the open-label extension (OLE) period and up to 57 weeks for participants entering the OLE period but not the long-term OLE.

The treatment duration will be up to 26 weeks for participants not entering the OLE period and up to 52 weeks for participants entering the OLE period but not the long-term OLE.

The number of visits will be up to 10 visits for participants not entering the OLE period and up to 16 visits for participants entering the OLE period but not the long-term OLE.

For participants who enter the long-term OLE, treatment and study participation will continue with visits every 12 weeks per protocol specifications.

ELIGIBILITY:
Inclusion Criteria:

* Participant ≥1 year post bilateral lung transplantation at the time of screening
* Participants presenting with CLAD Stage 1 or 2: FEV1 from >50% to 80% of post-transplant baseline at screening and at randomization
* Participants who have received at least 8 weeks of azithromycin (≥250 mg/day, at least 3 times a week) prior to randomization

Exclusion Criteria:

* FEV1 ≤50% of the post-transplant baseline value (CLAD 3 and 4)
* Lung function decline that can be explained by non-CLAD causes including but not limited to acute lung allograft rejection (>A1), antibody-mediated rejection, airway stenosis, or tracheobronchomalacia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-09-17 (Estimated); Study Completion 2028-06-02 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline to Week 26 in forced expiratory volume in 1 second (FEV1) | Baseline to Week 26

SECONDARY OUTCOMES:
Response rate at Week 26 | Baseline to Week 26
  Defined as the proportion of participants with ≤10% decline in FEV1 at Week 26 compared with baseline
Absolute change from baseline to Week 26 in FEV1 | Baseline to Week 26
Absolute change from baseline to Week 26 in percent predicted FEV1 | Baseline to Week 26
Percent change from baseline to Week 26 in forced vital capacity (FVC) | Baseline to Week 26
Absolute change from baseline to Week 26 in FVC | Baseline to Week 26
Absolute change from baseline to Week 26 in percent predicted FVC | Baseline to Week 26
Time to CLAD progression during the double-blind treatment period | Baseline to Week 26
  Defined as the first of the following events: >10% decline in FEV1 compared with baseline, or change in CLAD stage, or re-transplantation, or death
Time to re-transplantation or death | Up to 7 days after the administration of last dose of study drug
Percent change from baseline to Week 26 in 6-minute walk distance | Baseline to Week 26
Absolute change from baseline to Week 26 in 6-minute walk distance | Baseline to Week 26
Change from baseline to Week 26 in Saint George Respiratory Questionnaire (SGRQ) | Baseline to Week 26
  Total score and scores by domain
Change from baseline to Week 26 in EQ-5D-5L | Baseline to Week 26
  Visual analogue scale and individual dimensions
Change from baseline to Week 26 in Patient-Reported Outcomes Measurement Information System-29 profile version 2.1 | Baseline to Week 26
  Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29) profile V2.1 (domain scores)
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to 7 days after the administration of last dose of study drug
  Treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs), as well as laboratory abnormalities during the double-blind treatment period and the open-label extensions

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (80):
- United States (33):
  - UAB Lung Health Center- Site Number : 8400026, Birmingham, Alabama
  - St. Joseph's Hospital & Medical Center - Norton Thoracic Research Department- Site Number : 8400019, Phoenix, Arizona
  - David Geffen School of Medicine at UCLA- Site Number : 8400020, Los Angeles, California
  - Stanford Health Care - Center for Advance Lung Disease- Site Number : 8400008, Stanford, California
  - Mayo Clinic- Site Number : 8400031, Jacksonville, Florida
  - University of Miami - Jackson Memorial Hospital- Site Number : 8400030, Miami, Florida
  - Advent Health Transplant Institute- Site Number : 8400023, Orlando, Florida
  - Tampa General Hospital- Site Number : 8400015, Tampa, Florida
  - ~Emory University Hospital- Site Number : 8400027, Atlanta, Georgia
  - Northwestern University- Site Number : 8400003, Chicago, Illinois
  - Loyola University Medical Center- Site Number : 8400025, Maywood, Illinois
  - University Of Iowa Hospitals And Clinics- Site Number : 8400032, Iowa City, Iowa
  - University of Maryland School of Medicine- Site Number : 8400009, Baltimore, Maryland
  - ~Johns Hopkins University School of Medicine- Site Number : 8400034, Baltimore, Maryland
  - Brigham & Women's Hospital/VA Boston Lung Transplant Program- Site Number : 8400016, Boston, Massachusetts
  - University of Michigan Hospital - 1500 E Medical Center Dr- Site Number : 8400014, Ann Arbor, Michigan
  - Corewell Health- Site Number : 8400010, Grand Rapids, Michigan
  - NYU Langone Medical Center- Site Number : 8400001, New York, New York
  - Icahn School of Medicine at Mount Sinai- Site Number : 8400037, New York, New York
  - New York Presbyterian/Columbia University Medical Center- Site Number : 8400002, New York, New York
  - Montefiore Medical Center- Site Number : 8400036, The Bronx, New York
  - Duke Lung Transplant Program- Site Number : 8400017, Durham, North Carolina
  - Cleveland Clinic Foundation- Site Number : 8400005, Cleveland, Ohio
  - OSU Wexner Medical Center- Site Number : 8400028, Columbus, Ohio
  - University of Pennsylvania - Harron Lung Center- Site Number : 8400006, Philadelphia, Pennsylvania
  - Temple University Hospital- Site Number : 8400007, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center- Site Number : 8400018, Nashville, Tennessee
  - Baylor University Medical Center - Dallas- Site Number : 8400011, Dallas, Texas
  - UT Southwestern Medical Center- Site Number : 8400013, Dallas, Texas
  - Baylor University Medical Center - Houston- Site Number : 8400024, Houston, Texas
  - Houston Methodist Research Institute- Site Number : 8400021, Houston, Texas
  - UT Health San Antonio - University Hospital- Site Number : 8400035, San Antonio, Texas
  - Inova Fairfax Medical Campus - IHVI ALD and Lung Transplant Services- Site Number : 8400004, Falls Church, Virginia
- Australia (3):
  - Investigational Site Number : 0360003, Darlinghurst, New South Wales
  - Investigational Site Number : 0360001, Chermside, Queensland
  - Investigational Site Number : 0360002, Murdoch, Western Australia
- Investigational Site Number : 0400001, Vienna, Austria
- Belgium (2):
  - Investigational Site Number : 0560002, Godinne
  - Investigational Site Number : 0560001, Leuven
- Canada (3):
  - Investigational Site Number : 1240002, Edmonton, Alberta
  - Investigational Site Number : 1240001, Vancouver, British Columbia
  - Investigational Site Number : 1240004, Toronto, Ontario
- China (9):
  - Investigational Site Number : 1560004, Beijing
  - Investigational Site Number : 1560002, Chengdu
  - Investigational Site Number : 1560008, Fuzhou
  - Investigational Site Number : 1560007, Guangzhou
  - Investigational Site Number : 1560001, Hangzhou
  - Investigational Site Number : 1560005, Hefei
  - Investigational Site Number : 1560009, Shanghai
  - Investigational Site Number : 1560003, Wuxi
  - Investigational Site Number : 1560006, Zhengzhou
- Czechia (2):
  - Investigational Site Number : 2030002, Olomouc
  - Investigational Site Number : 2030001, Praha 5 - Motol
- Investigational Site Number : 2080001, Copenhagen, Denmark
- Investigational Site Number : 2460001, Helsinki, Finland
- France (6):
  - Investigational Site Number : 2500005, La Plessis Robinson
  - Investigational Site Number : 2500006, Marseille
  - Investigational Site Number : 2500004, Paris
  - Investigational Site Number : 2500002, Pessac
  - Investigational Site Number : 2500003, Saint-Herblain
  - Investigational Site Number : 2500001, Suresnes
- Investigational Site Number : 2760003, München, Germany
- Investigational Site Number : 3480001, Budapest, Hungary
- Investigational Site Number : 3760001, Petah Tikva, Israel
- Italy (5):
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico Milano-Site Number : 3800001, Milan, Milano
  - Investigational Site Number : 3800005, Padua
  - IRCCS-ISMETT (Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione)-Site Number : 3800004, Palermo
  - Fondazione IRCCS Policlinico San Matteo-Site Number : 3800003, Pavia
  - Azienda Ospedaliera Universitaria Senese UOC Malattie Respiratorie e Trapianto Polmonare-Site Number : 3800002, Siena
- Investigational Site Number : 5280001, Groningen, Netherlands
- Investigational Site Number : 5780001, Oslo, Norway
- South Korea (4):
  - Investigational Site Number : 4100004, Yangsan, Gyeongsangnam-do
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
- Spain (4):
  - Investigational Site Number : 7240002, A Coruña, A Coruña [La Coruña]
  - Investigational Site Number : 7240003, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240001, Santander, Cantabria
  - Investigational Site Number : 7240004, Valencia
- Investigational Site Number : 7520001, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17801 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25518&tenant=MT_SNY_9011